CLINICAL TRIAL: NCT04549311
Title: Perianal Abscess Recurrence and Fistula Formation: Antibiotics Following Incision and Drainage Trial - (PARFAIT) A Vanguard Randomized Controlled Trial
Brief Title: Perianal Abscess Recurrence and Fistula Formation: Antibiotics Following Incision and Drainage Trial
Acronym: PARFAIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Paul Karanicolas, Scientist and Associate Professor, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTO Project ID: 2122
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Perianal Abscess; Perianal Fistula
Keywords: Post-operative antibiotics
MeSH Terms: interventions — Amoxicillin; Clavulanic Acid; Ciprofloxacin; Metronidazole

STUDY DESIGN:
Intervention Model Description: Pragmatic, multicenter, open-label, three-arm parallel-group Vanguard feasibility randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antibiotic 1 arm (amoxicillin + clavulanic acid) (Active Comparator): Patients will undergo I&D of PA by the clinician as per standard of care. This may occur in the emergency department or operating room. Patients may or may not receive packing based on the clinician's standard practice and institutional routines.
  Patients randomized to the antibiotic 1 arm will receive a prescription for amoxicillin + clavulanic acid (875 mg amoxicillin and 125 mg clavulanic acid BID) PO for 7 days. Otherwise, all participants will be treated identically according to the institution's standard practices.
  Interventions: Drug: Antibiotic 1 arm (amoxicillin + clavulanic acid)
- Antibiotic 2 arm (ciprofloxacin + metronidazole) (Active Comparator): Patients will undergo I&D of PA by the clinician as per standard of care. This may occur in the emergency department or operating room. Patients may or may not receive packing based on the clinician's standard practice and institutional routines.
  Patients randomized to the antibiotic 2 arm will receive a prescription for ciprofloxacin + metronidazole (ciprofloxacin 500 mg and metronidazole 500 mg BID) PO for 7 days. Otherwise, all participants will be treated identically according to the institution's standard practices.
  Interventions: Drug: Antibiotic 2 arm (ciprofloxacin + metronidazole)
- No antibiotics (No Intervention): Patients will undergo I&D of PA by the clinician as per standard of care. This may occur in the emergency department or operating room. Patients may or may not receive packing based on the clinician's standard practice and institutional routines.
  In the comparator arm, patients will not receive any antibiotics. Otherwise, all participants will be treated identically according to the institution's standard practices.

INTERVENTIONS:
Drug: Antibiotic 1 arm (amoxicillin + clavulanic acid) — Prescription of antibiotics (amoxicillin + clavulanic acid) after incision and drainage of perianal abscess.
  Arms: Antibiotic 1 arm (amoxicillin + clavulanic acid)
Drug: Antibiotic 2 arm (ciprofloxacin + metronidazole) — Prescription of antibiotics (ciprofloxacin + metronidazole) after incision and drainage of perianal abscess.
  Arms: Antibiotic 2 arm (ciprofloxacin + metronidazole)

SUMMARY:
Most perianal abscesses (PA) result from an infection originating in anal crypts that extend into anal glands in the intersphincteric plane. Patients commonly present to the ER and usually require surgical intervention, which poses a burden on the healthcare system. If left undrained, a PA can expand into the adjacent tissues as well as progress to systemic infection. One of the major complications of PA are perianal fistulae; the creation of a tract between the anal canal and the perianal skin that is lined with granulation tissue or skin cells. Up to 1/3 of patients with a PA will develop a fistula; which occurs if a PA drains spontaneously through the perianal skin, and the infection becomes chronic. If this happens, surgical intervention is needed and abscesses may reoccur. Post incision and drainage (I&D) antibiotics in PA have been used to address complications but their use is still controversial and there are no specific recommendations on their use to prevent the formations of fistulae.

Recent findings from a systematic review (6 studies, N=817 patients) published in 2019 demonstrated that antibiotic use following I&D of PA was associated with a 36% lower odds of fistula formation, though the quality of the evidence was low.

As there are no established prophylactic treatments for fistulae, and because they are difficult to treat, further study of this simple intervention seems warranted. In this trial, adults with a PA requiring I&D will be randomly assigned to receive standard of care with antibiotics or standard of care without antibiotics after I&D. This trial will be conducted under the IMPACTS (Innovative, Multicentre, Patient-centred Approach to Clinical Trials in Surgery) program umbrella and will follow IMPACTS methodology. For the Vanguard trial, the aim is to determine the feasibility of conducting a definitive trial. Future outcomes of interest are incidence of fistula formation (defined as drainage of the perianal region at or after 2 months), need for re-intervention (i.e., any intervention on the perianal region), quality of life, healthcare utilization, healing time and mortality.

DETAILED DESCRIPTION:
The development of perianal abscesses is relatively common with an estimated incidence in the UK of 40 per 100,000 habitants (Canadian incidence unknown). It is uncertain if there is any benefit to using prophylactic antibiotics after incision and drainage of a perianal abscess in order to reduce the formation of fistulae, the need for re-intervention, health system costs, and healing time. Further research from high-quality RCTs is needed to establish a benefit, if any, for this practice.

Objectives: Before embarking on a definitive RCT, this pilot trial has five specific feasibility objectives:

1. To assess our ability to accrue patients using the IMPACTS Program design platform at multiple institutions, over the course of one year.
2. To assess our ability to adaptively randomize patients and deliver the randomized assignment using the IMPACTS Program design platform, over the course of one year.
3. To assess our ability to collect complete data directly from participants (patients and clinicians) on: re-intervention, fistula formation, quality of life, and healing time over the course of one year.
4. To examine our ability to carry out data linkages using the IMPACTS Program design platform over the course of one year.
5. To estimate the incidence of fistula formation to inform the sample size calculation for the definitive trial.

Study design: This is a multicentre, pragmatic, open label, three-arm parallel-group Vanguard feasibility randomized controlled trial. Adult patients with perianal abscesses requiring incision and drainage will be randomized to receive standard of care with antibiotics or standard of care without antibiotics after incision and drainage. If feasibility is demonstrated during the pilot trial, we will plan to conduct a definitive trial. If there are only minimal changes to the protocol, we will include data from the pilot phase into the definitive trial analysis (i.e. a Vanguard design).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Perianal abscess requiring incision and drainage

Exclusion Criteria:

* Allergies or contraindications to amoxicillin + clavulanic acid, penicillin, ciprofloxacin, or metronidazole
* Definite need to be on antibiotics at the treating clinicians' discretion
* Immunosuppression such as: human immunodeficiency virus (HIV), chronic steroids treatment, current chemotherapy
* Abscess associated with Inflammatory Bowel Disease (IBD)
* Supralevator perianal abscess
* Recurrent perianal abscesses within 5 years
* Known rectal cancer diagnosis within 5 years
* History of pelvic radiotherapy within 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-01-22 (Actual); Study Completion 2023-01-22 (Actual)

PRIMARY OUTCOMES:
Total number of participants accrued across all sites, per month | 1 year
  Feasible if 3 or more patients accrued per month between all sites
Proportion of participants who received the allocated intervention, across all sites | 1 year
  Feasible if >90% of patients receive correct intervention
Proportion of complete data collection for patient-reported outcome surveys, across all sites | 1 year
  Feasible if >80% of data is collected
Proportion of successful data linkage of patient-reported outcome data with Institute of Clinical Evaluative Sciences dataset(s) | 1 year
  Feasible if linkage is possible in >90% of patients
Estimation of fistula formation in three groups | 1 year
  Rate of fistula formation in the three groups

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karanicolas, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- Canada (3):
  - North York General Hospital, North York, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No